CLINICAL TRIAL: NCT05080400
Title: Effects of Gellan Gum on the Glycemic, Gastrointestinal and Appetitive Responses to a White Rice Meal Assessed by MRI
Brief Title: White Rice and Effect of Gellan Gum on Glucose Responses by MRI
Acronym: WIGG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Luca Marciani, Professor of Gastrointestinal Imaging, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 470-2001
Record Dates: First submitted 2021-08-11; First posted 2021-10-15 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Glycemic Response to Feeding in Healthy Participants
Keywords: white rice; glycemia; gellan gum; hydrocolloids
MeSH Terms: interventions — gellan gum

STUDY DESIGN:
Intervention Model Description: randomised 2-way crossover study
Who Masked: Participant
Masking Description: Participant blind to cooking process
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gellan gum (Experimental): White rice cooked with gellan gum
  Interventions: Dietary Supplement: White rice; Dietary Supplement: Gellan gum
- Control (Placebo Comparator): White rice cooked without gellan gum
  Interventions: Dietary Supplement: White rice

INTERVENTIONS:
Dietary Supplement: White rice — Jasmine rice 179g of cooked weight
Dietary Supplement: Gellan gum — Food grade hydrocolloid polysaccharide 5.5g dissolved in 356g cooking water containing 185g rice
  Arms: Gellan gum

SUMMARY:
Rice is a staple food for over half the world's population. High consumption of white rice has been linked with high obesity and increased risk for type 2 diabetes. However, it is still the favoured type of rice among consumers, contributing to the observed increasing trends in diet-related diseases in countries with high rice consumption. Controlling the properties of white rice products (e.g. reducing the glycaemic index and/or increasing satiety) with relatively simple interventions could contribute to producing foods with health-promoting digestibility profiles.

One way to reduce the glycaemic index of white rice is through processing. Addition of food thickeners (called hydrocolloid gums) has previously been shown to reduce the digestibility of foods.

This work will test the hypothesis that gellan gum is a simple way to manipulate the body's glucose response to a white rice which in turn will have health-promoting effects. MRI imaging will be used to monitor the gastrointestinal responses.

DETAILED DESCRIPTION:
Addition of hydrocolloids has previously been shown to reduce the digestibility of foods. Hydrocolloids are polysaccharides used to increase viscosity and gelatinization and have many other applications in the food industry. However, there is a lack of mechanistic understanding on how these hydrocolloids may act during digestion in the human body. Preliminary in-house data suggested that the addition of gellan gum to rice cooking may reduce digestibility rates though mechanisms yet to be understood. This work will test the hypothesis that gellan gum can be used to manipulate white rice product properties to enhance health-promoting glycaemic, gastrointestinal and satiety responses in healthy human participants.

Aims:

1. to collect pilot data on postprandial glucose levels of isoenergetic test meal made from rice and Gellan Gum 2 . to collect data on their gastric emptying and satiety. 3. to compare postprandial glucose levels, gastric emptying and satiety for the treatments 4. to explore relationships between glucose levels, gastric emptying and satiety.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 18.5 and ≤ 24.9 kg/m2
* Able to give informed consent
* Apparently healthy: no medical conditions or previous gastrointestinal surgery which might affect study measurements (judged by the investigators)

Exclusion Criteria:

* Fasting fingerprick screening blood sugar level higher than 5.4 mmol/L
* Restrained eating behaviour as determined by Eating habits and SCOFF screening questionnaires
* Not used to eating breakfast
* Not used to eating three meals a day
* Use of medication which interferes with study measurements for example acid suppressants or anti-spasmodics.
* Participation in another nutritional or biomedical trial 3 months before the pre-study screening or during the study.
* Reported participation in night shift work during the two weeks prior to pre-study investigation or during the study. Night work is defined as working between midnight and 6.00 AM.
* Strenuous exercise for more than10 hours per week.
* Consumption of ≥21 alcoholic drinks in a typical week
* Reported weight loss or gain ≥ 10 % of bodyweight during the six months period before the pre-study examination.
* Following a medically- or self-prescribed diet during the two weeks prior to the pre-study examination and until the end of the study
* Dislike of the products served as the dietary test treatments including the pasta meal
* Any allergy or food intolerance to the test treatments
* Not suitable for MRI scanning (e.g., presence of metal implants, infusion pumps and pacemakers) as assessed by standard MRI safety questionnaire.
* Pregnancy or breastfeeding declared by candidate
* Antibiotic or prescribed probiotic treatment in the past 12 weeks
* Inability to lie flat
* Poor understanding of the spoken and/or written English language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Incremental Area Under the Curve of post prandial blood glucose up to 2h (iAUC2h) | 2 hours
  Fingerprick blood glucose area under the curve for 2 hours

SECONDARY OUTCOMES:
Ad libitum objective pasta meal at the end of the study day | 3 hours
  Weighted amount of ad libitum pasta meal consumed at end of study morning
Under the Curve for appetite scores post prandial up to 2 hours (AUC2h) | 2 hours
  Area under the curve of Visual Analogue Scores up to 2 hours postprandially

OTHER OUTCOMES:
Time to Peak of blood glucose | 2 hours
  Fingerprick blood glucose time to peak
Peak blood glucose | 2 hours
  Fingerprick blood glucose peak value
Area Under the Curve of post prandial gastric volumes up to 2h (AUC2h) | 2 hours
  Gastric volumes area under the curve from MRI images
Visual appearance of meal in the stomach | 2 hours
  Descriptive intragastric appearance (e.g. layering, boluses) of meal in the stomach
Small bowel water content area under the curve (AUC2h) | 2 hours
  Area under the curve of volume of freely mobile water in the small bowel from MRI images
Explorative correlations | 2 hours
  Explorative correlations between Fingerprick blood glucose area under the curve for 2 hours, Gastric volumes area under the curve from MRI images up to 2 hours postprandially and Area under the curve of appetite Visual Analogue Scores up to 2 hours postprandially

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Digestive Disases Centre , University of Nottingham, Nottingham, United Kingdom